CLINICAL TRIAL: NCT07174375
Title: Efficacy and Safety of PCSK9 Inhibitors in Patients With Acute Ischemic Stroke Undergoing Endovascular Therapy: A Prospective, Multicenter, Open-Label, Parallel, Randomized Controlled Clinical Trial
Brief Title: PCSK9 Inhibitors in Acute Ischemic Stroke Patients Undergoing Endovascular Therapy
Acronym: PCSK9-PROVE
Status: Not yet recruiting | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Nanfang Hospital, Southern Medical University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NFEC-2025-213
Record Dates: First submitted 2025-09-12; First posted 2025-09-15 (Actual); Last update posted 2025-09-15 (Actual); Status verified 2025-09

CONDITIONS: Acute Ischemic Stroke
Keywords: acute ischemic stroke; endovascular therapy; PCSK9 inhibitors; Lipid-Lowering Therapy; Early Artery Reocclusion
MeSH Terms: conditions — Ischemic Stroke | interventions — evolocumab; alirocumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Standard therapy plus PCSK9 inhibitor (Experimental): Patients in the Standard therapy plus PCSK9 inhibitor group will receive a subcutaneous injection of either Evolocumab (420 mg) or Alirocumab (150 mg) within 48 hours after endovascular therapy, followed by subsequent subcutaneous injections of Evolocumab (420 mg) or Alirocumab (150 mg) every 4 weeks, for a total of 3 administrations.
  Interventions: Drug: PCSK9 inhibitor
- Standard therapy alone (No Intervention): Patients in the Standard therapy alone (control) group will receive standard of care treatment. If low-density lipoprotein cholesterol (LDL-C) levels fail to meet target goals after 7 days, cholesterol absorption inhibitors (e.g., Ezetimibe or Hypemab) may be administered. If LDL-C levels still remain suboptimal after 1 month, PCSK9 inhibitors may be added to the treatment regimen.

INTERVENTIONS:
Drug: PCSK9 inhibitor — PCSK9 (Proprotein Convertase Subtilisin/Kexin Type 9) inhibitors are a class of monoclonal antibody drugs that lower low-density lipoprotein cholesterol (LDL-C) by inhibiting the PCSK9 protein, which increases the liver's ability to remove LDL-C from the blood. This intervention involves the use of established PCSK9 inhibitor agents.
  Other Names: Evolocumab; Alirocumab
  Arms: Standard therapy plus PCSK9 inhibitor

SUMMARY:
This is a prospective, multicenter, randomized controlled clinical study to evaluate the efficacy of PCSK9 inhibitor in addition to standard therapy in patients with acute ischemic stroke undergoing endovascular therapy.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years.
* Meets the diagnostic criteria for acute ischemic stroke according to the Chinese Guidelines for the Diagnosis and Treatment of Acute Ischemic Stroke 2023.
* Severe stenosis or occlusion of large anterior circulation vessels confirmed by DSA, MRA, or CTA.
* Preoperative NIHSS score ≥ 4 and < 25.
* Meets the indications for endovascular therapy per the Chinese Guidelines for Endovascular Therapy of Acute Ischemic Stroke 2023, and successful reperfusion of the target vessel (mTICI ≥ 2b) achieved via emergency endovascular intervention.
* LDL-C > 1.8 mmol/L or non-HDL cholesterol > 2.6 mmol/L.
* Signed informed consent provided by the patient or their legally authorized representative.

Exclusion Criteria:

* Confirmed non-atherosclerotic causes of vascular stenosis/occlusion (e.g., cardioembolism, vasculitis, vascular malformation, moyamoya disease, iatrogenic causes).
* History of intracranial hemorrhage or systemic bleeding within the past 3 months.
* Presence of hemorrhagic transformation (PH1/PH2) immediately after the procedure.
* Severe hepatic impairment: ALT > 3 times the upper limit of normal, INR > 1.2, hepatic encephalopathy, or history of drug-induced liver injury.
* Use of PCSK9 inhibitors within 6 months prior to enrollment.
* Pre-stroke mRS ≥ 2.
* Terminal illness (e.g., malignancy, end-stage renal disease) with an expected survival of < 3 months.
* Pregnancy or lactation.
* Other neurological diseases that may interfere with neurological function assessment during follow-up.
* Allergy or intolerance to PCSK9 inhibitors or statins.
* Participation in another interventional clinical trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 478 (Estimated)
Dates: Start 2025-09-15 (Estimated); Primary Completion 2027-12-15 (Estimated); Study Completion 2027-12-15 (Estimated)

PRIMARY OUTCOMES:
Functional outcome: The proportion of mordified Rankin Scale of 0 to 2 points | 90 days after the stroke onset
  The proportion of mordified Rankin Scale of 0 to 2 points at 90 days

SECONDARY OUTCOMES:
Proportion of patients with early neurological improvement | 7 days post-treatment
  Defined as a reduction of ≥4 points on the National Institutes of Health Stroke Scale (NIHSS) score or a complete resolution of neurological deficits (NIHSS=0) within 7 days after treatment.
Incidence of target vessel reocclusion or recurrent infarction | 90 days after the stroke onset
  Reocclusion of the responsible vessel confirmed by CTA/MRA/DSA, or new cerebral infarction in the same territory confirmed by diffusion-weighted MRI.
Reduction amplitude of low-density lipoprotein (LDL-C) | Within 7 days post-treatment
  Absolute and relative reduction of LDL-C levels from baseline to Day 7.
Mortality rate | 90 days after the stroke onset
  All-cause mortality at 90 days.
Incidence of symptomatic hemorrhagic transformation | Within 7 days post-treatment
  Hemorrhagic transformation associated with neurological deterioration (increase in NIHSS ≥4 points) confirmed by CT or MRI.
Incidence of acute liver injury | Within 90 days post-treatment
  Alanine aminotransferase (ALT) or aspartate aminotransferase (AST) >3 times the upper limit of normal.
Proportion of patients with early neurological deterioration | Within 7 days post-treatment
  Defined as an increase of ≥4 points on the NIHSS score within 7 days post-treatment.
Distribution of modified Rankin Scale (mRS) scores | 90 days after the stroke onset
  Shift analysis of mRS scores at 90 days (range 0-6).
Incidence of malignant brain edema | 48 to 96 hours after onset
  Defined as the presence of cerebral edema with mass effect on cranial CT or MRI within 48 to 96 hours after symptom onset, including midline shift ≥ 5 mm and/or compression of ventricles or cisterns.
Midline shift distance | 72 to 96 hours after onset
  Maximum distance of midline shift (in millimeters) measured on axial CT or MRI.
Incidence of adverse events | Within 90 days post-treatment
  All adverse events and serious adverse events, recorded and graded according to CTCAE v5.0.

CONTACTS AND LOCATIONS:
Locations (12):
- China (12):
  - Fujian Medical University Union Hospital, Fuzhou, Fujian
  - Dongguan Donghua Hospital, Dongguan, Guangdong
  - Dongguan People's Hospital, Dongguan, Guangdong
  - Huadu District People's Hospital of Guangzhou, Guangzhou, Guangdong
  - Nanfang Hospital of Southern Medical University, Guangzhou, Guangdong
  - Heyuan People's Hospital, Heyuan, Guangdong
  - Hengzhou City People's Hospital, Guangxi, Hengzhou, Guangxi (Autonomous Region)
  - Hainan Provincial Hospital of Traditional Chinese Medicine, Haikou, Hainan
  - Haikou People's Hospital, Haikou, Hainan
  - Hainan Provincial People's Hospital, Haikou, Hainan
  - The Second Affiliated Hospital of Hainan Medical University, Haikou, Hainan
  - Ganzhou City People's Hospital, Ganzhou, Jiangxi

IPD SHARING:
Plan to Share IPD: No